CLINICAL TRIAL: NCT06662279
Title: Hyrax Vs. Invisalign Palatal Expander Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Align Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A025375
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Malocclusions; Narrow Maxilla; Narrow Maxillary Arch; Crowding
MeSH Terms: conditions — Malocclusion; Crowding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Invisalign Palatal Expander (Active Comparator)
  Interventions: Device: Removable Rapid Palatal Expander
- Hyrax Expander (Active Comparator)
  Interventions: Device: Banded Palatal Expander

INTERVENTIONS:
Device: Removable Rapid Palatal Expander — Removable palatal expander where expanders are changed to obtain up to .25mm expansion per expander
  Arms: Invisalign Palatal Expander
Device: Banded Palatal Expander — Palatal expander cemented into mouth where a screw is turned to obtain .25mm expansion per turn
  Arms: Hyrax Expander

SUMMARY:
The purpose of this study is to compare expansion result and the overall experience between the Invisalign Palatal Expander and the Hyrax expander.

ELIGIBILITY:
Inclusion Criteria:

* Subject ages 6-11 years old
* Subject must need maxillary expansion
* Subjects must have erupted dentition in the area of the primary molars or permanent premolars and the first permanent molar

Exclusion Criteria:

* Subjects with palatal exostosis/surface aberration/ cleft palate
* Subject's dentition not compatible with device or allergy to device materials
* Subject with active caries, periodontal disease, TMD

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
width of palate after expansion | from enrollment to study completion, approximately 4 months
  intraoral scans will be taken of the subject's upper arch, including palate throughout the study and widths will be measured

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orange Coast Orthodontics, Laguna Hills, California
  - Spillers Orthodontics, Warner Robins, Georgia
  - Innovative Orthodontic Centers, Naperville, Illinois
  - The Orthodontic Studio, Chevy Chase, Maryland